CLINICAL TRIAL: NCT01316692
Title: A Phase II Correlative Clinical Trial of MLN8237, a Selective Aurora Kinase A (AURKA) Inhibitor, in Patients With Unresectable Stage III or Stage IV Melanoma Disease
Brief Title: Aurora A Kinase Inhibitor MLN8237 in Treating Patients With Unresectable Stage III-IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine; Director, Melanoma and Tumor Immunotherapy, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC MEL 1036; NCI-2010-02322 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01FD003522 (FDA)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Recurrent Melanoma; Stage IIIc Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Biopsy; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MLN8237 (Experimental): Patients receive oral Aurora A kinase inhibitor MLN8237 every 12 hours on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker identification and analysis; Procedure: biopsy; Other: immunohistochemistry/tissue microarrays; Genetic: TdT-mediated dUTP nick end labeling assay; Other: mass spectrometry

INTERVENTIONS:
Other: laboratory biomarker identification and analysis — Correlative studies
  Other Names: protein expresssion analysis
Procedure: biopsy — Correlative studies
  Other Names: selective tissue excision
Other: immunohistochemistry/tissue microarrays — Correlative studies
Genetic: TdT-mediated dUTP nick end labeling assay — Correlative studies
  Other Names: TUNEL assay
Other: mass spectrometry — Correlative studies

SUMMARY:
RATIONALE: Aurora A kinase inhibitor MLN8237 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well Aurora A kinase inhibitor MLN8237 works in treating patients with unresectable stage III-IV melanoma

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the degree of clinical benefit based primarily on objective clinical responses with AURKA inhibitor, MLN8237 in patients with metastatic melanoma in a phase II, 2-stage trial for patients with measurable unresectable disease.

SECONDARY OBJECTIVES:

I. Assess the progression-free survival and overall survival for all patients enrolled.

II. Define toxicities due to MLN8237 and characterize their severity both over a short and prolonged duration of administration.

III. In patients entered on stage 1 of clinical trial whenever possible through pre-treatment biopsy and post-treatment surgical specimen, we will define target inhibition at tumor sites based on: AURKA autophosphorylation (AURKAThr288/AURKA), intra-tumoral drug levels, expression of p53-induced NOXA and PUMA expression, TPX2, (by IHC) and TUNEL as markers of apoptosis, cell cycle changes (mitotic index), proliferation (Ki-67), aneuploidy, and AKT phosphorylation.

IV. All phase II trial patients enrolled on the 2nd stage will have pre- and post-treatment biopsies (post-day 7+/-3 days) to demonstrate that AURKA is inhibited based on autophosphorylation AURKA/AURKA^Thr 288, Histone H3 (at S10) phosphorylation, AKT phosphorylation, cell cycle changes (mitotic index), TPX2 (by IHC), proliferation (Ki-67), aneuploidy, and p53-induced NOXA and PUMA expression, and TUNEL as markers of apoptosis.

V. Demonstrate any correlation between MLN8237 induced target inhibition at tumor sites and clinical benefit of MLN8237.

VI. Characterize the de novo molecular mutational profile of the melanomas from all patients entered using a developed SNaPshot assay for melanoma in addition loss of regulatory proteins (i.e., PTEN), DNA copy numbers and gene expression (AURKA), and autophosphorylation of AURKA as well as AURKA localization by IHC.

OUTLINE: Patients receive oral Aurora A kinase inhibitor MLN8237 every 12 hours on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIc or IV histologically proven melanoma (confirmed by Vanderbilt pathologists), that is not curable by standard surgery, radiation therapy, or chemotherapy. No available effective therapy (i.e.; therapy known to be curative,). Non-biopsied (resected) tumor sites must be measurable for therapy.
* Patients on stage 2 of the enrollment must have tumor sites that are easily biopsied and be willing to undergo pre- and post-treatment (around day 8 +/- 3 days) tumor biopsies.
* Adequate performance status for the study, ECOG 0-1
* Adequate baseline organ system function, including

  1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 without growth factor support
  2. Hemoglobin ≥ 9.0g/dL (without need for transfusion support within 30 days; growth factor allowed)
  3. Platelet count ≥100,000 cells/mm3 without transfusion or growth factor requirement
  4. INR<1.5,
  5. Creatinine < 1.5x institutional upper limit of normal (IULN), and/or an adequate renal function as defined by: Calculated creatinine clearance must be ≥ 40 mL/minute (Cockcroft-Gault).
  6. Aspartate and alanine aminotransferase < 2.5 x institutional upper limit of normal (IULN), bilirubin < 1.5x IULN
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 3 months after the completion of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study and for 3 months after the completion of the study
* A single regimen of prior chemotherapy for metastatic melanoma is allowed. Patients also may have received other immunotherapy or biologic therapy (including kinase inhibitors, antibodies to checkpoints CTLA4, PD1, PDL1, etc.) for metastatic melanoma and there is a limit of three therapy regimens
* No prior Aurora kinase inhibitor
* Completed prior chemotherapy a minimum of 4 weeks previously (6 weeks for BCNU and/or mitomycin C), 4 weeks for prior immune therapy, 6 weeks for antibodies to checkpoints CTLA4, PD1, PDL1, etc, and 2 weeks for targeted agents (i.e. inhibitors of MEK, BRAF, Akt, PI3K, mTORC1/2) or localized radiation therapy. All treatment All treatment related toxicity must have resolved to grade 2 or less or to a baseline level as well.
* Patients cannot receive concomitant radiation therapy at enrollment. While on protocol limited palliative radiotherapy extending over a small bone marrow field (10%) is allowed.
* Patients with brain metastases are allowed only if they are off systemic corticosteroids and stable for a minimum of 8 weeks.
* Patients must be 18 years of age or above and voluntary written informed consent must be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Subject must be able to take oral medication and to maintain a fast as required before and after MLN8237 administration.

Exclusion Criteria

* Uncontrolled or serious infection
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patients with thromboembolic disease cannot be on coumadin, but low molecular heparins are allowed.
* Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
* Prior allogeneic bone marrow or organ transplantation.
* Concurrent therapy for cancer.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Inability to comply with protocol-specified procedures (i.e., treatment, monitoring, or follow-up)
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patients with GI absorptive problems making it unlikely to absorb study medication or more likely to experience GI toxicities.
* Patient is HIV-positive and is receiving combination antiretroviral therapy.
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study
* Other serious medical problem that in the view of the investigator makes therapy difficult to comply with or difficult to interpret toxicity
* If applicable, patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has received other investigational drugs with 14 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sosman, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants on this study were treated at Vanderbilt-Ingram Cancer Center. The study was conducted from October 2011- August 2015
Pre-assignment Details: A total of 19 patients consented to participate in this study. Four of 19 patients were screen failures and therefore were not eligible, 3 patients were eligible, but withdrew before treatment.
Period: Overall Study
Arm/Group | MLN8237
Started | 12
Completed | 0
Not Completed | 12
Not completed — Adverse Event | 5
Not completed — Disease Progression | 7

BASELINE CHARACTERISTICS:
Arm/Group | MLN8237
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: If 2 or more of 23 pts show CR/PR in stage 1, then an additional 33 pts will be enrolled in stage 2. If 6 or more of the total 56 pts show CR/PR at 18 weeks, then further clinical trials will be warranted. Per Response Evaluation Criteria in Solid Tumor (RECIST)1.1: Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: At 18 weeks
Population: All patients with Objective Response, defined as a complete or partial response.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | MLN8237
Number analyzed (Participants) | 12
participants | 0 [0 to 0.265]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the duration in time from start of therapy to last follow-up, disease progression, or death for any reason.measured every 6 weeks for 24 weeks, and then every 12 weeks or to last date known alive or death, determined every 6 months for up to 5 years. For those who are alive and without progression, they are censored at the last date known alive.
Time Frame: On treatment date to last follow-up, disease progression or death for any reason, up to 5 years
Population: All patients are included in the analysis on intention-to treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MLN8237
Number analyzed (Participants) | 12
days | 111 [45 to 187]

3. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details) Evaluated every 3 months for 12 months, then every 6 months
Time Frame: On treatment date to last follow-up or death for any reason, up to 5 years
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MLN8237
Number analyzed (Participants) | 12
days | 256 [136 to 419]

4. Secondary Outcome: Number of Grade 3 and 4 Study-related Toxicities
Description: Event are graded using National Cancer Institute Common Toxicity Criteria with grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening/disabling, 5 = death. toxicities measured on day 1 of each 21-day cycle. Treatment continues to disease progression, toxicity, or withdrawal for other reasons.
Time Frame: at 18 weeks
Population: total numbers of adverse events, patients experiencing grade 3 and 4 related to study treatment
Measure: Number; unit: toxicities
Arm/Group | MLN8237
Number analyzed (Participants) | 12
toxicities
  Grade 3 Toxicities | 6
  Grade 4 Toxicities | 3
  Grade 5 Toxicities1 | 0

5. Other Pre Specified Outcome: Characterize the de Novo Molecular Mutation Profile of the Melanomas for Association Between Objective Responses to MLN8237 in Patients With Pre-treatment Melanoma Tissue.
Description: In stage 1 patients: tumor biopsies are taken before initiation of treatment and on the 8th day of the first cycle of treatment. Tissue will be assayed for mutations that are neither parent-possessed, nor able to be transmitted, in pre- and in post-treatment tissue and the results will be compared and contrasted with patients' objective clinical responses, as determined by RECIST 1.1, after 18 weeks of treatment
Time Frame: At 24 weeks
Population: Collected samples of tumors were very limited. It did not allow us to perform the described assays
Arm/Group | MLN8237
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Correlation Between MLN8237-induced Selective Aurora Kinase A Inhibition in Post-treatment Tumor Sites and Clinical Benefit of MLN8237
Description: In stage 2 patients: tumor biopsies are taken before initiation of treatment and on the 8th day of the first cycle of treatment. Post-treatment tumor tissue will be assayed for MLN8237-induced selective Aurora Kinase A inhibition and compared to pre-treatment tumor tissue and the results will be compared and contrasted with patients' objective clinical responses, as determined by RECIST 1.1, after 18 weeks of treatment
Time Frame: At 24 weeks
Population: unable to collected the required number of tumor samples
Arm/Group | MLN8237
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years, 10 months
Arm/Group | MLN8237
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN8237 (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial infection (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN8237 (N=12)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (17)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (10)
Mucositis oral (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 6 (9)
Vomiting (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (12)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 8 (11)
Chills (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
administration site conditions (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (14)
White blood cell decreased (Investigations) | 6 (12)
Neutrophil count decreased (Investigations) | 5 (9)
Platelet count decreased (Investigations) | 3 (9)
Alkaline phosphatase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 7 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes